CLINICAL TRIAL: NCT07223762
Title: Hyperangulated Versus Standard Geometry Laryngoscope Blade Trial
Acronym: ANGLE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Casey, Primary Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 250433
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure
Keywords: critical illness; emergency airway management; tracheal intubation; video laryngoscope
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Parallel group, pragmatic, randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperangulated video laryngoscope blade (Active Comparator): For patients assigned to the hyperangulated video laryngoscope blade group, the operator will use a hyperangulated video laryngoscope blade on the first laryngoscopy attempt.
  Interventions: Other: Hyperangulated video laryngoscope blade
- Standard Geometry Video Laryngoscope Blade Group (Active Comparator): For patients assigned to the standard geometry laryngoscope blade group, the operator will use a standard geometry video laryngoscope blade on the first laryngoscopy attempt.
  Interventions: Other: Standard geometry video laryngoscope blade

INTERVENTIONS:
Other: Hyperangulated video laryngoscope blade — Hyperangulated video laryngoscope blade
  Arms: Hyperangulated video laryngoscope blade
Other: Standard geometry video laryngoscope blade — Standard geometry video laryngoscope blade
  Arms: Standard Geometry Video Laryngoscope Blade Group

SUMMARY:
The Hyperangulated versus Standard Geometry Laryngoscope Blade (ANGLE) Trial is a multi-center, non-blinded, parallel-group, randomized clinical trial evaluating the effect of use of a hyperangulated video laryngoscope blade versus use of a standard geometry video laryngoscope blade. Critically ill adults undergoing tracheal intubation in participating EDs and ICUs who meet eligibility criteria will be enrolled and randomly assigned in a 1:1 ratio to either intubation using a hyperangulated video laryngoscope blade or a standard geometry video laryngoscope blade. The primary outcome is the incidence of successful intubation on the first attempt. The secondary outcome is incidence of hypoxemia during the interval between induction and 2 minutes after tracheal intubation.

DETAILED DESCRIPTION:
Clinicians frequently perform tracheal intubation of critically ill patients in the emergency department (ED) or intensive care unit (ICU). In 10-20% of emergency tracheal intubations, clinicians are unable to intubate the trachea on the first attempt, which increases the risk of complications during intubation. To intubate the trachea, clinicians use a device called a laryngoscope, which consists of a handle with an attached blade. Clinicians intubate by holding the laryngoscope handle and inserting the blade into the patient's mouth to (1) visualize the opening to the trachea (the larynx) and (2) create a pathway through which an endotracheal tube can be advanced through the oropharynx and larynx and into the trachea.

Video laryngoscopes use a camera embedded in the laryngoscope blade to transmit images of the airway to a screen that can be viewed in real time by the clinician to aid endotracheal tube placement. Video laryngoscopes have been shown to improve the ability of clinicians to view the larynx and increase the likelihood of successful intubation on the first attempt, compared to direct laryngoscopes, which do not have a camera or a screen. A recent multicenter randomized trial found that, among 1,417 adults undergoing tracheal intubation in an ED or ICU, the incidence of successful intubation on the first attempt was 85% with a video laryngoscope and 70% with a direct laryngoscope (absolute difference, 14.3; 95% CI, 9.9 to 18.7). Use of a video laryngoscope is now standard of care for tracheal intubation in many EDs and ICUs and is recommended in international guidelines.

Two types of laryngoscope blades are available for use with video laryngoscopes in clinical care. Standard geometry video laryngoscope blades were designed to approximate the shape of Macintosh direct laryngoscopes, the preferred tool before the advent of video laryngoscopy. When using a standard geometry laryngoscope blade, the clinician inserts the blade into the mouth, displaces the tongue, and lifts up and away from the operator to elevate the epiglottis and expose the vocal cords. Because this approach creates a direct line-of-site view of the vocal cords, the clinician may view the vocal cords directly (with the naked eye) or indirectly on the video screen. Creating this line-of-site view of the vocal cords with a standard angulation blade may require more effort than with a hyperangulated blade, but it creates a direct pathway for passage of an endotracheal tube through the mouth and into the trachea. Because use of a standard geometry laryngoscope blade includes creation of a direct pathway for passage of an endotracheal tube, some experts have hypothesized that use of a standard geometry laryngoscope blade could increase the incidence of successful intubation on the first attempt, compared to use of hyperangulated blades.

Hyperangulated video laryngoscope blades were designed to have a more acute angle that more closely matches the natural curvature of the airway, allowing a view of the vocal cords with less manipulation of the airway. Because use of a hyperangulated blade does not include creation of a direct, line-of-sight view of the vocal cords, it is only used for indirect laryngoscopy with a video laryngoscope. When using a hyperangulated video laryngoscope blade, the clinician inserts the hyperangulated blade into the mouth, displaces the tongue, and then gently tilts the blade to view the vocal cords. While use of a hyperangulated blade may make it easier to obtain a view of the vocal cords, the pathway for passage of an endotracheal tube through the mouth and into the trachea may be less direct than with a standard geometry video laryngoscope blade. Some experts have hypothesized that, by making it easier to obtain a view of the vocal cords, use of a hyperangulated video laryngoscope blade may increase the incidence of successful intubation on the first attempt, compared to use of a standard geometry video laryngoscope blade.

Two randomized controlled trials among adults intubated by anesthesiologists during elective tracheal intubation in the operating room reported different effects of use of a hyperangulated versus standard geometry video laryngoscope blade on the incidence of successful intubation on the first attempt. Köhl et al reported a 30% increase in the incidence of successful intubation on the first attempt with use of a hyperangulated video laryngoscope blade (97% vs 67%; p=0.002) in patients with anticipated difficult airways. In contrast, Zhang et al reported a non-significant increase in the incidence of successful intubation on the first attempt with use of a standard geometry video laryngoscope blade (79% vs 71%; p=0.26) in patients in cervical immobilization.

Emergency tracheal intubation in the ED and ICU differs significantly from elective tracheal intubation in the operating room. Patients are more likely to have difficult airway characteristics that might make it more challenging to obtain a complete view of the larynx (e.g., cervical spine immobilization during trauma), rates of failure on the first attempt and complications during intubation are significantly higher, and clinicians performing intubation have less prior experience performing intubation, on average. No prior randomized trials have compared hyperangulated blades to standard geometry blades during intubation using a video laryngoscope in the ED or ICU. To determine the effect of use of a hyperangulated video laryngoscope blade versus a standard geometry video laryngoscope blade on the incidence of successful intubation on the first attempt among critically ill adults undergoing intubation in the ED or ICU, a randomized trial is needed.

ELIGIBILITY:
Inclusion Criteria

1. Patient is located in a participating unit.
2. Planned procedure is orotracheal intubation using a laryngoscope.
3. Planned operator is a clinician expected to routinely perform tracheal intubation in the participating unit.

Exclusion Criteria:

1. Patient is known to be less than 18 years old.
2. Patient is known to be pregnant.
3. Patient is known to be a prisoner.
4. Immediate need for tracheal intubation precludes safe performance of study procedures.
5. Operator has determined that use of a direct laryngoscope is required for the optimal care of the patient.
6. Operator has determined that use of a hyperangulated video laryngoscope blade or a standard geometry video laryngoscope blade is required or contraindicated for the optimal care of the patient either because of factors related to the patient (e.g., patient's upper airway anatomy requires a specific blade type) or the operator (e.g., treating clinicians lack sufficient comfort with one of the blade types).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Successful intubation on the first attempt. | Duration of placement of the endotracheal tube, an average duration of two minutes.
  Successful intubation on the first attempt is defined as placement of an endotracheal tube in the trachea with a single insertion of a laryngoscope blade into the mouth and EITHER a single insertion of an endotracheal tube into the mouth OR a single insertion of a bougie into the mouth followed by a single insertion of an endotracheal tube over the bougie into the mouth.

SECONDARY OUTCOMES:
Hypoxemia | During the interval between induction and 2 minutes after tracheal intubation.
  The secondary outcome is hypoxemia, defined as a peripheral oxygen saturation < 85% during the interval between induction and 2 minutes after tracheal intubation.

OTHER OUTCOMES:
Cormack-Lehane grade of glottic view | Duration of placement of the endotracheal tube, an average duration of two minutes.
  Cormack-Lehane grade of glottic view on the first laryngoscopy attempt
Number of laryngoscopy attempts | Duration of placement of the endotracheal tube, an average duration of two minutes.
Number of bougie attempts | Duration of placement of the endotracheal tube, an average duration of two minutes.
Number of endotracheal tube attempts | Duration of placement of the endotracheal tube, an average duration of two minutes.
Duration of intubation | Duration of placement of the endotracheal tube, an average duration of two minutes.
  The time (in seconds) between the initial insertion of the laryngoscope blade into the mouth and the final placement of an endotracheal tube or tracheostomy tube in the trachea.
Severe complications during intubation | Between induction and 2 minutes after intubation.
  The development of one or more of the following between induction and 2 minutes after intubation: (1) severe hypoxemia (SpO2 <80%), (2) severe hypotension (systolic blood pressure <80 mm Hg or new or increased vasopressor administration), and (3) cardiac arrest.
Esophageal intubation | Duration of placement of the endotracheal tube, an average duration of two minutes.
Injury to the teeth | Duration of placement of the endotracheal tube, an average duration of two minutes.
Operator-reported aspiration | Duration of placement of the endotracheal tube, an average duration of two minutes.
In-hospital death by 1 hour | 1 hour
In-hospital death by 28 days | In the first 28 days after enrollment
Ventilator-free days through day 28 | In the first 28 days after enrollment
ICU-free days through day 28 | In the first 28 days after enrollment

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado, Denver Anschutz Medical Campus, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Our Lady of the Lake Hospital, Inc., Baton Rouge, Louisiana
  - Ochsner Clinic Foundation, Jefferson, Louisiana
  - University of Maryland Baltimore, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Zhang J, Tan LZ, Toh H, Foo CW, Wijeratne S, Hu H, Seet E. Comparing the first-attempt tracheal intubation success of the hyperangulated McGrath(R) X-blade vs the Macintosh-type CMAC videolaryngoscope in patients with cervical immobilization: a two-centre randomized controlled trial. J Clin Monit Comput. 2022 Aug;36(4):1139-1145. doi: 10.1007/s10877-021-00746-5. Epub 2021 Aug 4. PMID 34347225
- [Result] Kohl V, Wunsch VA, Muller MC, Sasu PB, Dohrmann T, Peters T, Tolkmitt J, Dankert A, Krause L, Zollner C, Petzoldt M. Hyperangulated vs. Macintosh videolaryngoscopy in adults with anticipated difficult airway management: a randomised controlled trial. Anaesthesia. 2024 Sep;79(9):957-966. doi: 10.1111/anae.16326. Epub 2024 May 24. PMID 38789407
- [Result] Paik H, Park HP. Randomized crossover trial comparing cervical spine motion during tracheal intubation with a Macintosh laryngoscope versus a C-MAC D-blade videolaryngoscope in a simulated immobilized cervical spine. BMC Anesthesiol. 2020 Aug 15;20(1):201. doi: 10.1186/s12871-020-01118-3. PMID 32799791
- [Result] Suppan L, Tramer MR, Niquille M, Grosgurin O, Marti C. Alternative intubation techniques vs Macintosh laryngoscopy in patients with cervical spine immobilization: systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2016 Jan;116(1):27-36. doi: 10.1093/bja/aev205. Epub 2015 Jun 30. PMID 26133898
- [Result] van Zundert A, Pieters B, Doerges V, Gatt S. Videolaryngoscopy allows a better view of the pharynx and larynx than classic laryngoscopy. Br J Anaesth. 2012 Dec;109(6):1014-5. doi: 10.1093/bja/aes418. No abstract available. PMID 23154957
- [Result] Kleine-Brueggeney M, Greif R, Schoettker P, Savoldelli GL, Nabecker S, Theiler LG. Evaluation of six videolaryngoscopes in 720 patients with a simulated difficult airway: a multicentre randomized controlled trial. Br J Anaesth. 2016 May;116(5):670-9. doi: 10.1093/bja/aew058. PMID 27106971
- [Result] Hansel J, Rogers AM, Lewis SR, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adults undergoing tracheal intubation. Cochrane Database Syst Rev. 2022 Apr 4;4(4):CD011136. doi: 10.1002/14651858.CD011136.pub3. PMID 35373840
- [Result] Prekker ME, Driver BE, Trent SA, Resnick-Ault D, Seitz KP, Russell DW, Gaillard JP, Latimer AJ, Ghamande SA, Gibbs KW, Vonderhaar DJ, Whitson MR, Barnes CR, Walco JP, Douglas IS, Krishnamoorthy V, Dagan A, Bastman JJ, Lloyd BD, Gandotra S, Goranson JK, Mitchell SH, White HD, Palakshappa JA, Espinera A, Page DB, Joffe A, Hansen SJ, Hughes CG, George T, Herbert JT, Shapiro NI, Schauer SG, Long BJ, Imhoff B, Wang L, Rhoads JP, Womack KN, Janz DR, Self WH, Rice TW, Ginde AA, Casey JD, Semler MW; DEVICE Investigators and the Pragmatic Critical Care Research Group. Video versus Direct Laryngoscopy for Tracheal Intubation of Critically Ill Adults. N Engl J Med. 2023 Aug 3;389(5):418-429. doi: 10.1056/NEJMoa2301601. Epub 2023 Jun 16. PMID 37326325
- [Result] Prekker ME, Trent SA, Lofrano A, Russell DW, Barnes CR, Brewer JM, Doerschug KC, Gaillard JP, Gandotra S, Ginde AA, Ghamande S, Gibbs KW, Hughes CG, Janz DR, Khan A, Mitchell SH, Page DB, Rice TW, Self WH, Smith LM, Stempek SB, Vonderhaar DJ, West JR, Whitson MR, Casey JD, Semler MW, Driver BE. Laryngoscopy and Tracheal Intubation: Does Use of a Video Laryngoscope Facilitate Both Steps of the Procedure? Ann Emerg Med. 2023 Oct;82(4):425-431. doi: 10.1016/j.annemergmed.2023.02.016. Epub 2023 Apr 5. PMID 37028995
- [Result] Park L, Zeng I, Brainard A. Systematic review and meta-analysis of first-pass success rates in emergency department intubation: Creating a benchmark for emergency airway care. Emerg Med Australas. 2017 Feb;29(1):40-47. doi: 10.1111/1742-6723.12704. Epub 2016 Oct 27. PMID 27785883
- [Result] Brown CA 3rd, Bair AE, Pallin DJ, Walls RM; NEAR III Investigators. Techniques, success, and adverse events of emergency department adult intubations. Ann Emerg Med. 2015 Apr;65(4):363-370.e1. doi: 10.1016/j.annemergmed.2014.10.036. Epub 2014 Dec 20. PMID 25533140
- [Result] Russotto V, Myatra SN, Laffey JG, Tassistro E, Antolini L, Bauer P, Lascarrou JB, Szuldrzynski K, Camporota L, Pelosi P, Sorbello M, Higgs A, Greif R, Putensen C, Agvald-Ohman C, Chalkias A, Bokums K, Brewster D, Rossi E, Fumagalli R, Pesenti A, Foti G, Bellani G; INTUBE Study Investigators. Intubation Practices and Adverse Peri-intubation Events in Critically Ill Patients From 29 Countries. JAMA. 2021 Mar 23;325(12):1164-1172. doi: 10.1001/jama.2021.1727. PMID 33755076
- [Result] Law JA, Duggan LV, Asselin M, Baker P, Crosby E, Downey A, Hung OR, Kovacs G, Lemay F, Noppens R, Parotto M, Preston R, Sowers N, Sparrow K, Turkstra TP, Wong DT, Jones PM; Canadian Airway Focus Group. Canadian Airway Focus Group updated consensus-based recommendations for management of the difficult airway: part 2. Planning and implementing safe management of the patient with an anticipated difficult airway. Can J Anaesth. 2021 Sep;68(9):1405-1436. doi: 10.1007/s12630-021-02008-z. Epub 2021 Jun 8. PMID 34105065
- [Result] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475